Title: The causal relationship between serum vitamin D level

and hepatitis B virus replication in patients with chronic

hepatitis B virus infection

NCT 03068767

Date of document: 1, June 2017

IRB approval letter (as attached)

**Statistical Analyses Plan** 

Statistical analysis was performed using SPSS version 16.0 (SPSS Inc. Chicago, IL).

Data were analyzed by chi-square test and student's t test. The correlation among

serum vitamin D and FIB-4 was analyzed using Pearson's correlation analysis. The

significance in all of the tests was two-tailed and a p value of less than 0.05 was